CLINICAL TRIAL: NCT01872442
Title: Combination of Dasatinib and Peg-Interferon Alpha 2b in First Line for Chronic Myeloid Leukemia in Chronic Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DASA-PegIFN
Record Dates: First submitted 2013-05-14; First posted 2013-06-07 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Phase of Chronic Myeloid Leukemia
MeSH Terms: interventions — Dasatinib; peginterferon alfa-2b

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasatinib (Experimental): Dasatinib,Bristol Myers Squibb
  Interventions: Drug: Dasatinib; Drug: Peg-Interferon alpha2b
- Peg-Interferon alpha2b (Experimental): Peg-Interferon alpha2b (Peg-IFN α2b), Merck
  Interventions: Drug: Dasatinib; Drug: Peg-Interferon alpha2b

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 100mg daily starting at inclusion
  If ANC ≤ 1.5.109/L, platelets ≤ 100.0.109/L or lymphocytes > 4.0.109/L at 3 months, dasatinib will be continued alone, and patients will be still followed in the study
Drug: Peg-Interferon alpha2b — 30 µg weekly starting month 4- month 21

SUMMARY:
Interferon alpha was a therapy used in Chronic Myeloid Leukemia in Chronic phase prior to the advent of tyrosine kinase inhibitors. Synergistic effect of the combination of Peg-IFNα2a with Imatinib was demonstrated in the clinical SPIRIT trial. In this study, the investigators address the question of the efficacy and safety of dasatinib in combination with low dose of Peg-IFNα-2b as frontline therapy for patients with newly diagnosed Chronic Myeloid Leukemia in Chronic phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent.
2. Target Population

   a)18 to 65 years b)Newly diagnosed (≤ 3 months) Philadelphia chromosome positive chronic CP-CML c)Major BCR-ABL transcripts d)Not previously treated for CML except with hydroxyurea or anagrelide e)ECOG Performance Status≤ 2 f)Adequate Organ Function. i)Total bilirubin< 2.0 times the institutional Upper Limit of Normal ii)Hepatic enzymes(AST, ALT )≤ 2.5 ULN iii)Serum Na, K+, Mg2+ and Ca2+ > Lower Limit of Normal (LLN) or supplemented iv)Serum Creatinine< 1.5 ULN g)Women of childbearing potential (WOCBP) must be using an adequate method of contraception.
3. Free subject, without guardianship nor subordination,
4. Health insurance coverage. -

Exclusion Criteria:

1. Patients with BCR-ABL other than M-BCR-ABL, Philadelphia negative CML.
2. Patients previously treated with Tyrosine Kinase Inhibitors (TKIs).
3. Medical history and concurrent diseases :

   1. Hypersensitivity to any of the excipients of dasatinib
   2. Prior treatment with Interferon-α, contraindication to interferon-α, hypersensitivity to any of the excipients of PegIFNα2b,
   3. Concomitant immunosuppressive treatment or corticosteroids,
   4. Preexisting thyroid disease unless it is controlled with conventional treatment, Auto-immune thyroiditis,
   5. Autoimmune disorder, Chronic liver disease,
   6. Prior or ongoing severe psychiatric disease,
   7. Epilepsy or compromised central nervous system(CNS) function,
   8. HIV positivity, chronic hepatitis B or C,
   9. Uncontrolled or significant cardio vascular or pulmonary disease,

   i)Uncontrolled angina, myocardial infarction or congestive heart failure within 6 months, ii)Echocardiography with LVF < 45% or LLN, peak velocity of tricuspid regurgitant flow > 2,8 m/s iii)Pulmonary arterial hypertension (PAH), iv)Any history of clinically significant ventricular or supraventricular arrhythmias, v)Diagnosed congenital long QT syndrome, vi)Prolonged QTc interval > 450 msec (Fredericia) on 3 pre-entry electrocardiogram, vii)Subjects with hypokalemia or hypomagnesemia if it cannot be corrected, j)Other malignant disease during the last 5 years prior to the inclusion except basal cell carcinoma of the skin or carcinoma in situ of the cervix, k)History of significant bleeding disorder unrelated to CML, including: i)Diagnosed congenital bleeding disorders (e.g. von Willebrand's disease), ii)Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding. l)Another severe or life -threatening medical disease.
4. Women who are pregnant or breastfeeding, WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after the last dose of study drug.
5. Prohibited treatments and/or therapies:

   1. strong inhibitors of the CYP3A4,
   2. category I drugs that are generally accepted to have a risk of causing "Torsades de Pointes", Patients must discontinue the drug minimum 7 days prior to starting dasatinib.
6. History /any condition for poor compliance to the treatment.
7. Inability to freely provide consent through judiciary or administrative condition.
8. Ongoing participation to another study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-10-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of molecular response | at 12 months.
  Molecular response 4.5 (MR4.5) is defined by either a positive BCR-ABL/ABL ratio ≤ 0.0032 on the international scale or by undetectable BCR-ABL with the analysis of at least 32000 copies of ABL (according to the ELN recommendations by N. Cross et al., leukemia 2012).
  Centralized analyses of molecular response by RTQPCR will be performed for all molecular assessments in this study.

SECONDARY OUTCOMES:
Rate of complete cytogenetic response | 3, 6, 12, 18, 24 months, and every 12 months thereafter.
Rate of major molecular responses | 3, 6, 9, 12, 15, 18, 21, 24 months and every 6 months thereafter.
Rate of molecular response | 6, 9, 12, 15, 18, 21, 24 months and every 6 months thereafter.
  Rate of molecular response 4.5 and 5.0
Kinetics and duration | 6, 9, 12, 15, 18, 21, 24 months and every 6 months thereafter
  Cumulative rate, Kinetics and duration CCR, MMR, MR4.5, MR5.0
Rate of PegIFN-α2b and dasatinib discontinuation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lydia ROY, MD, Principal Investigator — Poitiers University Hospital

REFERENCES:
- [Derived] Roy L, Chomel JC, Guilhot J, Guerci-Bresler A, Escoffre-Barbe M, Giraudier S, Charbonnier A, Dubruille V, Huguet F, Johnson-Ansah H, Lenain P, Ame S, Etienne G, Nicolini FE, Rea D, Cony-Makhoul P, Courby S, Ianotto JC, Legros L, Machet A, Coiteux V, Hermet E, Cayssials E, Bouchet S, Mahon FX, Rousselot P, Guilhot F; French CML Group (FiLMC). Dasatinib plus Peg-Interferon alpha 2b combination in newly diagnosed chronic phase chronic myeloid leukaemia: Results of a multicenter phase 2 study (DASA-PegIFN study). Br J Haematol. 2023 Jan;200(2):175-186. doi: 10.1111/bjh.18486. Epub 2022 Oct 10. PMID 36214090